CLINICAL TRIAL: NCT05664308
Title: Single-center Pilot Study to Evaluate the Interest of a Hybrid Connected Watch for Heart Rate Monitoring in Postoperative Cardiac Surgery
Brief Title: Interest of a Hybrid Connected Watch for Cardiac Rhythm Monitoring in Post-operative Cardiac Surgery
Acronym: MONHYCARD
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0604
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation
Keywords: Post Operative Atrial Fibrillation; Connected Watch
MeSH Terms: conditions — Atrial Fibrillation | interventions — epicatechin gallate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Electrocardiogram
  Interventions: Other: Clinical follow-up (ECG)
- Electrocardiogram + Connect Watch
  Interventions: Other: Clinical follow-up (ECG); Other: Ongoing monitoring

INTERVENTIONS:
Other: Clinical follow-up (ECG) — Clinical follow-up with a consultation at the University Hospital at 3, 6, and 12 months, with an ECG at each visit.
Other: Ongoing monitoring — Once operated, patients will be monitored remotely via a computerized data transfer routine anonymized by the WITHINGS software, based on the data from the watch.
  It's contractually agreed with WITHINGS that the transmissions will be scheduled and transmitted weekly to the center.
  Groups: Electrocardiogram + Connect Watch

SUMMARY:
The objective of this single-center pilot study is, with the help of a connected watch, to show the absence of recurrence or maintenance of sinus rhythm in patients with a Post Operative Atrial Fibrillation (POAF) and to help treating cardiologists in the care of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Major with an indication for conventional cardiac surgery with de novo postoperative AF onset.
* Agreeing to participate in the study and having signed an informed consent.
* Agreeing to undergo 12 months of postoperative monitoring.

Exclusion Criteria:

* Patient with pre-operative AF
* Patient who does not have a smartphone compatible with the connected watch.
* Patient unable to perform an ECG measurement independently.
* Patient with a physical constraint to the measurement (arteriovenous fistula...)
* Minors
* Pregnant or breast-feeding women
* Adults under guardianship, under curatorship
* Patients whose life expectancy is less than 1 year
* Patients participating in another therapeutic trial likely to impact the evaluation criteria of the MONHYCARD study
* Contraindication to long-term anticoagulants
* Patients implanted with a mechanical valve prosthesis pre-operatively or after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with postoperative atrial fibrillation meeting the study eligibility criteria
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2028-03-19 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of recurrence of paroxysmal or persistent atrial fibrillation with continuous 12-month postoperative cardiac surgery monitoring in patients with POAF versus traditional follow-up with ECG recording at 3, 6 and 12 months | 12 months
  Recurrence rate of paroxysmal or persistent Atrial Fibrillation (AF) (ESC 2020 Definition) over a 12-month follow-up period post cardiac surgery according to traditional ECG monitoring at 3, 6, and 12 months more or less combined with connected watch monitoring

SECONDARY OUTCOMES:
Assessment of the rate of patients on anticoagulant therapy by follow-up modality | 12 months
  Rate of anticoagulant use at 3, 6, and 12 months according to rhythm status in both modalities
Evaluation of complication rates related to the different treatments according to the follow-up modality | 12 months
  Cardiovascular mortality, ischemic stroke, anticoagulant-related events
Assessment of the number of patients in AF | 12 months
  Postoperative AF rate in each group
Assessment of the duration of AF transitions | 12 months
  Postoperative AF rate over periods of more than 6 hours and/or 12 hours
Assessment of quality of life and satisfaction with use by follow-up modality | 12 months
  European Quality of Life-5 Dimensions (EQ-5D), (the maximum value is 3 (wich is the worse outcome) and the minimum is 1 (wich is the best outcome)), before intervention, at 3, 6 and 12 months
Assessment of quality of life and satisfaction with use by follow-up modality | 12 months
  Hospital Anxiety and Depression scale (HAD) scores, (the maximum value is 21 (wich is the worse outcome) and the minimum is 0 (wich is the best outcome)), before intervention, at 3, 6 and 12 months
Evaluate the appropriateness of each of the two modalities with treating cardiologists | 12 months
  Satisfaction questionnaire for treating cardiologists

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided